CLINICAL TRIAL: NCT00001242
Title: Studies of States With Resistance to Vitamin D and Parathyroid Hormone
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 890173; 89-DK-0173
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Hypocalcemia; Pseudohypoparathyroidism; Osteomalacia; Rickets; Pseudopseudohpoparathyroidism
Keywords: Rickets; Hypocalcemia; Albright Hereditary Osteodystrophy; Pseudohypoaldosteronism; Natural History
MeSH Terms: conditions — Hypocalcemia; Pseudohypoparathyroidism; Osteomalacia; Rickets; Pseudohypoaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Study Cohort: Patients of any age or sex with vitamin D resistance, rickets, osteomalacia, pseudohypoparathyroidism, pseudo- pseudohypoparathyroidism, or suspicion of these or related disorders

SUMMARY:
Patients with confirmed or suspected states with resistance to vitamin D or parathyroid hormone (PTH) will be admitted for diagnosis, treatment review with suggestions for modifications to the current or new treatment and for inclusion in other protocols. These states include hypocalcemia, rickets, osteomalacia, pseudohypoparathyroidism. Resistance to a factor is manifested by deficient bioeffect despite high levels of the factor in blood. Patients will be tested with multiple indices of mineral metabolism to establish the diagnosis and examine the spectrum of the underlying disorder. The principal therapies will be combinations of calcium, phosphate, and a vitamin D analog. Selected patients will have localization and surgery to remove a tumor that causes renal wasting of phosphate. Patients will also be considered for entry into other research protocols.

DETAILED DESCRIPTION:
Patients with confirmed or suspected states with resistance to vitamin D or parathyroid hormone (PTH) will be admitted for diagnosis, treatment review with suggestions for modifications to the current or new treatment and for inclusion in other protocols. These states include hypocalcemia, rickets, osteomalacia, pseudohypoparathyroidism. Resistance to a factor is manifested by deficient bioeffect despite high levels of the factor in blood. Patients will be tested with multiple indices of mineral metabolism to establish the diagnosis and examine the spectrum of the underlying disorder. The principal therapies will be combinations of calcium, phosphate, and a vitamin D analog. Selected patients will have localization and surgery to remove a tumor that causes renal wasting of phosphate. Patients will also be considered for entry into other research protocols.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients, from 2 months to 100 years of age, of either sex M or F, with vitamin D resistance, rickets, osteomalacia, pseudohypoparathyroidism, pseudo-pseudohypoparathyroidism, or suspicion of these or related disorders based upon the appropriateness of their problem to ongoing investigations.

Current investigations are focused principally upon the inclusion of subjects with, or suspected of having, hypocalcemia likely due to a resistance to parathyroid hormone, including subjects who have a diagnosis, or likely diagnosis, of pseudohypoparathyroidism or pseudopseudohypoparathyroidism.

Ages: 2 Months to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed or suspected states with resistance to vitamin D or parathyroid hormone (PTH)
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 1997-08-12 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
This study will provide information about problems relating to calcium in the blood, urine, and bones | take one to two weeks
  This is a natural history protocol, directed at diagnosing and managing the general clinical features in these patients. In addition the full clinical expression of certain rare disorders (target resistance to 1,25(OH)2D, pseudohypoparathyroidism, and pseudo- pseudohypoparathyroidism) will be characterized further. Some of these patients or their relatives will be entered into additional protocols, where appropriate for example, protocols to characterize the molecular causes of these disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Lee S Weinstein, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Marx SJ, Swart EG Jr, Hamstra AJ, DeLuca HF. Normal intrauterine development of the fetus of a woman receiving extraordinarily high doses of 1,25-dihydroxyvitamin D3. J Clin Endocrinol Metab. 1980 Nov;51(5):1138-42. doi: 10.1210/jcem-51-5-1138. PMID 6893458
- [Background] Nemeth AJ, Eaglstein WH, Falanga V, Hevia O, Taylor JR. Methods to speed healing after skin biopsy or trichloroacetic acid chemical peel. Prog Clin Biol Res. 1991;365:267-77. No abstract available. PMID 1862138
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1989-DK-0173.html